CLINICAL TRIAL: NCT04473859
Title: A Phase 1, Double-blind, Single Center, Controlled Study to Evaluate the Safety and Tolerability of FSR Peptide Versus Placebo Following Punch Biopsy in Adult Healthy Volunteers
Brief Title: Study to Evaluate the Safety of FSR Peptide Versus Placebo Following Punch Biopsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xequel Bio, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT1-01
Record Dates: First submitted 2020-07-10; First posted 2020-07-16 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Wound Heal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- FSR Peptide 20 μM (Experimental): Each subject will have two punch biopsies. FSR peptide will be applied to one punch biopsy. Placebo will be applied to the second punch biopsy.
  Interventions: Drug: FSR Peptide 20μM; Drug: Placebo
- FSR peptide 50 μM (Experimental): Each subject will have two punch biopsies. FSR peptide will be applied to one punch biopsy. Placebo will be applied to the second punch biopsy.
  Interventions: Drug: FSR Peptide 50μM; Drug: Placebo
- FSR peptide 100 μM (Experimental): Each subject will have two punch biopsies. FSR peptide will be applied to one punch biopsy. Placebo will be applied to the second punch biopsy.
  Interventions: Drug: FSR Peptide 100μM; Drug: Placebo
- FSR peptide 200 μM (Experimental): Each subject will have two punch biopsies. FSR peptide will be applied to one punch biopsy. Placebo will be applied to the second punch biopsy.
  Interventions: Drug: FSR Peptide 200μM; Drug: Placebo
- Placebo only (Placebo Comparator): Each subject will have two punch biopsies. Placebo will be applied to both punch biopsies.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FSR Peptide 20μM — Administered immediately after punch-biopsy and 24 hours after punch biopsy.
  Arms: FSR Peptide 20 μM
Drug: FSR Peptide 50μM — Administered immediately after punch-biopsy and 24 hours after punch biopsy.
  Arms: FSR peptide 50 μM
Drug: FSR Peptide 100μM — Administered immediately after punch-biopsy and 24 hours after punch biopsy.
  Arms: FSR peptide 100 μM
Drug: FSR Peptide 200μM — Administered immediately after punch-biopsy and 24 hours after punch biopsy.
  Arms: FSR peptide 200 μM
Drug: Placebo — Administered immediately after punch-biopsy and 24 hours after punch biopsy.

SUMMARY:
The purposes of this study is to test the safety of the study drug (FSR peptide) after a punch biopsy in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy subjects, 18-45 years of age and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* Female subjects must have been surgically sterilized at least six months prior to screening. Surgical sterilization procedures must be supported with clinical documentation made available to the sponsor and noted in the Relevant Medical History / Current Medical Conditions section of the CRF. OR: Postmenopausal women must have no regular menstrual bleeding for at least two years prior to inclusion. Menopause was to be confirmed by a plasma 17β-estradiol concentration of <20 pg/mL and a plasma FSH level of >40 IU/L.
* Normal sitting blood pressure and pulse rate , i.e.: BP: 100 - 140 mm Hg systolic, 50 - 90 mm Hg diastolic and pulse rate: 45 - 100 bpm. Blood pressure and pulse were to be measured after 3 minutes resting in a sitting position.
* Subject body mass index between 18 and 30 kg/m2
* Ability to communicate well with the investigator and comply with the requirements of the entire study.
* The subject has given his written consent to participate in the study.

Exclusion Criteria:

* History of serious adverse reactions or hypersensitivity to any drug.
* Presence or history of any allergy requiring acute or chronic treatment (seasonal) allergic rhinitis which requires no treatment may be tolerated).
* History of alcohol or drug abuse in the last 3 years.
* Abnormal physical findings of clinical significance at the screening examination or baseline which would interfere with the objectives of the study.
* Need of any prescription medication within 14 days prior to the administration of the drug and/or nonprescription medication within 7 days prior to the administration of the drug or anticipated need for any concomitant medication during the study.
* Participation in a clinical trial during the previous 4 weeks, i.e. from completion of the previous trial to the planned first administration of the current trial.
* Loss of 500 ml blood or more during the 3 month period before the study, e.g. as a donor.
* Existence of any surgical or medical condition which might interfere with the distribution, metabolism or excretion of the drug, i.e. impaired renal or hepatic function, diabetes mellitus, cardiovascular abnormalities, chronic symptoms of pronounced constipation or diarrhea or conditions associated with total or partial obstruction of the urinary tract.

Symptoms of a significant somatic or mental illness in the two week period preceding drug administration.

* History of hepatitis B and / or C and / or positive serology results which indicate the presence of hepatitis B and / or C.
* Positive results from the HIV serology.
* Clinically significant abnormal laboratory values (as determined by the Principal Investigator) at the screening evaluation. Serum albumin below 3.5 g/l (Note to File no. 8 states that the correct albumin value is below 35g/l) precludes study inclusion in any case.
* History of serious mental disorders.
* Positive results of the drug screening.
* History or clinical evidence of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurologic or other disease.
* Presence of any active skin pathology including e.g., acne, acute sunburn, inflammatory skin disease.
* Presence of any open wounds or infection on the same arm.
* History of skin disorders e.g. atopic eczema or psoriasis or keloid reaction(s) Any condition that constitutes a contraindication to minor surgical procedures (such as bleeding disorders) or that obliges to the use of prophylactic antibiotics (such as mitral valve prolapse) or other comedications for the performance of minor surgical procedures.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2008-03-06 (Actual); Primary Completion 2009-04-28 (Actual); Study Completion 2009-04-28 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events | Time of consent to day 28

SECONDARY OUTCOMES:
Time to healing | Up to 28 days
  The wound was clinically evaluated as healed or not healed.
Presence of hypertrophic granulation tissue | Up to 28 days
  Clinically assessed as present or not present. To qualify as present, there should be at least 3 mm granulation tissue protruding above the edge of the wound at any point of its perimeter.
Clinical General Impression scale on the evolution of the wound. | Up to 28 days
  Scale of 1-5: 1- Very bad; 2- Bad; 3- Fair; 4- Good; 5- Very Good
Wound height | day 28
  Assessed using the abbreviated Vancouver Scar Scale. The resulting abbreviated score was as follows. Scores are combined to calculate the final score.
  Pigmentation 0- Normal. Color that closely resembles the color over the rest of the subject's body
  1. Hypopigmentation
  2. Hyperpigmentation
  Vascularity 0- Normal. Color that closely resembles the color over the rest of the subject's body
  1. Pink
  2. Red
  3. Purple
Wound pliability | day 28
  Assessed using the abbreviated Vancouver Scar Scale. The resulting abbreviated score was as follows. Scores are combined to calculate the final score.
  Pigmentation 0- Normal. Color that closely resembles the color over the rest of the subject's body
  1. Hypopigmentation
  2. Hyperpigmentation
  Vascularity 0- Normal. Color that closely resembles the color over the rest of the subject's body
  1. Pink
  2. Red
  3. Purple
Histopathological evaluation of the area of the scar tissue | day 28
  Performed in a punch biopsy taken from the initial wound site at the end of the 28 day evaluation period.
Histopathological evaluation of the epidermal involution | day 28
  Performed in a punch biopsy taken from the initial wound site at the end of the 28 day evaluation period.
Histopathological evaluation of the rete pegs | day 28
  Performed in a punch biopsy taken from the initial wound site at the end of the 28 day evaluation period.
Histopathological evaluation of the area of granulation tissue | day 28
  Performed in a punch biopsy taken from the initial wound site at the end of the 28 day evaluation period.

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Ghatnekar, Principal Investigator — CEO
Locations (1):
- Swiss Pharma Contract Ltd, Allschwil, Switzerland